CLINICAL TRIAL: NCT00437658
Title: A Phase II, Randomized, Double-blind, Active-controlled Study to Assess the Safety and Efficacy of NBI-56418 in Subjects With Endometriosis
Brief Title: Elagolix Versus Subcutaneous Depot Medroxyprogesterone Acetate for the Treatment of Endometriosis
Acronym: PETAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-56418-0603
Record Dates: First submitted 2007-02-16; First posted 2007-02-21 (Estimated); Results first posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-03

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — elagolix; Medroxyprogesterone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Elagolix 75 mg BID (Experimental): Participants received elagolix 75 mg orally twice a day (BID) for 24 weeks and placebo to DMPA-SC by subcutaneous injection at weeks 1 and 12.
  Interventions: Drug: Elagolix; Drug: Placebo to DMPA-SC
- Elagolix 150 mg QD (Experimental): Participants received elagolix 150 mg orally once a day (QD) for 24 weeks and placebo to DMPA-SC by subcutaneous injection at weeks 1 and 12.
  Interventions: Drug: Elagolix; Drug: Placebo to DMPA-SC
- DMPA-SC (Active Comparator): Participants received placebo to elagolix orally once a day for 24 weeks and DMPA-SC 104 mg by subcutaneous injection at weeks 1 and 12.
  Interventions: Drug: Subcutaneous depot medroxyprogesterone acetate (DMPA-SC); Drug: Placebo to Elagolix

INTERVENTIONS:
Drug: Elagolix — Provided as tablets for oral administration
  Other Names: NBI-56418; Orilissa™
  Arms: Elagolix 150 mg QD; Elagolix 75 mg BID
Drug: Subcutaneous depot medroxyprogesterone acetate (DMPA-SC) — Provided for subcutaneous injection in a prefilled syringe, 104 mg/0.65 mL per syringe.
  Other Names: depo-subQ provera 104™
  Arms: DMPA-SC
Drug: Placebo to Elagolix — Matching placebo tablets for oral administration
  Arms: DMPA-SC
Drug: Placebo to DMPA-SC — Matching placebo for subcutaneous injection in a pre-filled syringe
  Arms: Elagolix 150 mg QD; Elagolix 75 mg BID

SUMMARY:
This study is designed to assess the effects of elagolix versus subcutaneous depot medroxyprogesterone acetate (DMPA-SC; also known as depo-provera) on bone mineral density (BMD) during treatment for 24 weeks with a subsequent 24-week post-treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Be female, aged 18 to 49 years, inclusive
* Have a total CPSSS of ≥ 6 at screening and baseline (Day 1) in the following categories: dysmenorrhea, dyspareunia, nonmenstrual pelvic pain, pelvic tenderness and induration. The total score must include a total of at least 2 in each of the categories of dysmenorrhea and nonmenstrual pelvic pain.
* Have had a diagnosis of endometriosis made following laparoscopic visualization of the disease within 8 years of the start of screening with recurrent or persistent symptoms.
* Have documented negative mammogram results within 12 months of screening if over the age of 40 years.
* Have menstrual cycles (28 days ±5 days). Assessment of cycle duration should be based on observations in the absence of drugs or conditions that are known to affect the cycle (e.g., oral contraceptives, leuprolide, pregnancy).
* Have a Body Mass Index (BMI) between 18 and 36 kg/m², inclusive.
* Agree to use two forms of nonhormonal contraception (e.g. condom with spermicide) during the study.

Exclusion Criteria:

* Are currently receiving gonadotropin-releasing hormone (GnRH) agonist, GnRH antagonist, danazol, or have received any of these agents within 6 months of the start of screening.
* Are currently receiving subcutaneous medroxyprogesterone acetate (DMPA-SC) or intramuscular medroxyprogesterone acetate (DMPA-IM) or have received any of these agents within 3 months of the start of screening.
* Have been nonresponsive to GnRH agonist or antagonist therapy for the management of endometriosis.
* Are currently using hormonal contraception or other forms of hormonal therapy or received such treatment within 1 month of the start of screening.
* Have had surgical treatment for endometriosis (laparoscopy) within 1 month of the start of screening.
* Have had a hysterectomy or bilateral oophorectomy.
* Have had prior treatment with NBI-56418.
* Have uterine fibroids or other pelvic lesions ≥ 5 cm in diameter
* Have any of the following abnormal cervical smear results at screening (based on the 2001 Bethesda System):

  * Benign endometrial cells (BEC) present, provided subject has irregular uterine bleeding or is over 40 years old
  * Atypical squamous cells of undetermined significance (ASC-US) present, and human papilloma virus (HPV) reflex testing is positive for high risk types or the testing outcome is unknown
  * Atypical squamous cells present, and high-grade squamous intraepithelial lesion (ASC-H) cannot be excluded
  * Atypical glandular cells of uncertain significance (AGUS/AGC): not otherwise specified (NOS), favor neoplasia (FN), favor endocervical, or favor endometrial origin types
  * Low-grade squamous intraepithelial lesion (LSIL) present
  * High-grade squamous intraepithelial lesion (HSIL) present
  * Adenocarcinoma in situ (AIS) / malignant cells present
* Have BMD with either lumbar spine or femur T-scores below -1.5 at screening as determined by the central DXA facility or have history of pathologic or compression fractures.
* Have been pregnant within 6 months of screening or currently breast feeding
* Are using systemic steroids on a chronic or regular basis within 3 months
* Have unstable medical condition or chronic disease
* Have chronic pelvic pain that is not caused by endometriosis

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 252 (Actual)
Dates: Start 2006-12-11 (Actual); Primary Completion 2008-11-24 (Actual); Study Completion 2008-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized at 58 centers in the United States.
Pre-assignment Details: This study consisted of a 24-week treatment period and a 24-week post-treatment period. Participants were randomized in a 1:1:1 ratio to one of three treatment groups.
Period: Treatment Period (24 Weeks)
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Started | 84 | 84 | 84
Received Study Drug | 84 | 84 | 84
Completed | 56 | 62 | 51
Not Completed | 28 | 22 | 33
Not completed — Adverse Event | 4 | 7 | 14
Not completed — Non-compliance | 1 | 1 | 4
Not completed — Withdrawal by Subject | 9 | 7 | 7
Not completed — Lack of Efficacy | 4 | 2 | 3
Not completed — Lost to Follow-up | 5 | 4 | 5
Not completed — Sponsor/Investigator Decision | 5 | 1 | 0
Period: Post-treatment Period (24 Weeks)
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Started | 56 | 62 | 51
Completed | 32 | 54 | 37
Not Completed | 24 | 8 | 14
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Non-compliance | 3 | 0 | 1
Not completed — Withdrawal by Subject | 12 | 6 | 8
Not completed — Lack of Efficacy | 0 | 2 | 2
Not completed — Lost to Follow-up | 5 | 0 | 1
Not completed — Sponsor/Investigator Decision | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC | Total
Number analyzed (Participants) | 84 | 84 | 84 | 252
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (7.5) | 31.4 (6.1) | 30.9 (6.3) | 31.6 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 84 | 84 | 252
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1 | 2
  Black | 6 | 10 | 10 | 26
  White | 68 | 70 | 65 | 203
  Hispanic | 8 | 4 | 6 | 18
  American Indian or Alaska Native, Caucasian | 0 | 0 | 1 | 1
  Black, Caucasian | 1 | 0 | 0 | 1
  Caucasian, Hispanic | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Bone Mineral Density of the Spine at Week 24
Description: Bone mineral density (BMD) was measured by dual X-ray absorptiometry (DXA). The percent change from baseline in spine and femur BMD at week 24 was assessed using a one-way analysis of variance (ANOVA) model. The absence of significant bone loss was supported if the lower bounds of the confidence intervals for the mean percent change in BMD were ≥ -2.2% for both the spine and femur at week 24.
Time Frame: Baseline and week 24
Population: Participants who received at least one dose (i.e., one tablet or injection) of study drug (safety analysis set) with available BMD data at both time points
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 55 | 62 | 50
percent change | -0.11 [-0.70 to 0.48] | -1.29 [-1.85 to -0.74] | -0.99 [-1.61 to -0.37]

2. Primary Outcome: Percent Change From Baseline in Bone Mineral Density of the Femur at Week 24
Description: as for outcome 1
Time Frame: Baseline and week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 56 | 64 | 51
percent change | -0.47 [-0.96 to 0.02] | -1.02 [-1.48 to -0.56] | -1.29 [-1.80 to -0.77]

3. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density of the Spine at Weeks 12 and 48
Description: Bone mineral density (BMD) was measured by dual X-ray absorptiometry (DXA). The percent change from baseline in BMD was assessed using a one-way analysis of variance (ANOVA) model.
Time Frame: Baseline and weeks 12 and 48
Population: Participants who received at least one dose (i.e., one tablet or injection) of study drug (safety analysis set) with available BMD data at each time point
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 84
percent change
  Week 12: number analyzed (Participants) | 68 | 68 | 67
  Week 12 | -0.39 [-0.80 to 0.02] | -1.05 [-1.46 to -0.64] | -0.57 [-0.98 to -0.15]
  Week 48: number analyzed (Participants) | 34 | 56 | 40
  Week 48 | 0.20 [-0.57 to 0.96] | -0.49 [-1.09 to 0.10] | -0.56 [-1.27 to 0.15]

4. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density of the Femur at Weeks 12 and 48
Description: as for outcome 3
Time Frame: Baseline and weeks 12 and 48
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 84
percent change
  Week 12: number analyzed (Participants) | 67 | 70 | 68
  Week 12 | -0.63 [-1.02 to -0.24] | -0.54 [-0.92 to -0.17] | -0.77 [-1.16 to -0.39]
  Week 48: number analyzed (Participants) | 33 | 57 | 39
  Week 48 | -0.38 [-1.10 to 0.33] | -0.86 [-1.41 to -0.32] | -0.76 [-1.42 to -0.10]

5. Secondary Outcome: Change From Baseline in N-telopeptide at Weeks 12, 24 and 48
Description: Blood samples to determine N-telopeptide concentrations were analyzed by a central laboratory using an enzyme-linked immunosorbent assay (ELISA). Change from baseline in N-telopeptide was analyzed using a one-way ANOVA model.
Time Frame: Baseline and weeks 12, 24 and 48
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: nM bone collagen equivalents (BCE)
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 84
nM bone collagen equivalents (BCE)
  Week 12: number analyzed (Participants) | 70 | 68 | 63
  Week 12 | 0.94 (0.43) | 0.57 (0.43) | 0.74 (0.45)
  Week 24: number analyzed (Participants) | 57 | 61 | 49
  Week 24 | 0.23 (0.50) | -0.30 (0.48) | -0.24 (0.54)
  Week 48: number analyzed (Participants) | 33 | 52 | 36
  Week 48 | -1.28 (0.61) | -1.53 (0.48) | -1.39 (0.58)

6. Secondary Outcome: Percentage of Participants With a Response in the Dysmenorrhea Component of the Composite Pelvic Signs and Symptoms Score (CPSSS) at Week 24
Description: The CPSSS consists of 5 components that address dysmenorrhea (pain during menstruation), dyspareunia (painful intercourse), non-menstrual pelvic pain, pelvic tenderness, and pelvic induration (hardening). Each component was scored on a scale of 0 to 3 (0 = absent, 1 = mild, 2 = moderate, and 3 = severe). The dysmenorrhea score was based on the participant's response to the question "Have you had painful menstruation during the last 28 days?".
  Participants were classified as responders for dysmenorrhea if they reported a 1 point or greater reduction (improvement) from baseline.
Time Frame: Baseline and week 24
Population: All randomized participants who received at least one oral dose of study drug, an initial subcutaneous injection, and either reported at least 7 e-diary visual analog scale (VAS) values or provided an assessment of either dysmenorrhea or non-menstrual pelvic pain at week 4 or later during the treatment phase (intent-to-treat) with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 57 | 65 | 51
percentage of participants | 86.0 | 73.8 | 86.3
Statistical Analysis 1: Comparison: Elagolix 150 mg QD vs DMPA-SC; Test type: Non-Inferiority — Statistical non-inferiority was defined when the lower bound of the 95% 2-sided confidence interval for the difference between an elagolix dose and DMPA-SC in the response rate was no less than -20% at week 24 for both dysmenorrhea and non-menstrual pelvic pain; p = 0.9630, Pearson chi-squared; Difference in response rates = -0.3, 95% CI 2-sided [-13.4 to 12.7] — Difference in response rate = elogolix - DMPA-SC
Statistical Analysis 2: Comparison: Elagolix 75 mg BID vs DMPA-SC; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p = 0.1010, Pearson chi-squared; Difference in response rates = -12.4, 95% CI 2-sided [-26.7 to 1.8] — Difference in response rate = elogolix - DMPA-SC

7. Secondary Outcome: Percentage of Participants With a Response in the Non-menstrual Pelvic Pain Component of the CPSSS at Week 24
Description: The CPSSS consists of 5 components that address dysmenorrhea, dyspareunia, non-menstrual pelvic pain, pelvic tenderness, and pelvic induration. Each component was scored on a scale of 0 to 3 (0 = absent, 1 = mild, 2 = moderate, and 3 = severe). The non-menstrual pelvic pain score was based on participant's response to the question "Have you had pelvic pain during the last 28 days?" Participants were classified as responders for non-menstrual pelvic pain if they reported a 1 point or greater reduction (improvement) from baseline.
Time Frame: Baseline and week 24
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 57 | 65 | 51
percentage of participants | 86.0 | 76.9 | 76.5
Statistical Analysis 1: Comparison: Elagolix 150 mg QD vs DMPA-SC; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p = 0.2048, Pearson chi-squared; Difference in response rates = 9.5, 95% CI 2-sided [-5.2 to 24.2] — Difference in response rates = elagolix - DMPA-SC
Statistical Analysis 2: Comparison: Elagolix 75 mg BID vs DMPA-SC; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p = 0.9544, Pearson chi-squared; Difference in response rates = 0.5, 95% CI 2-sided [-15.1 to 16.0] — Difference in response rates = elagolix - DMPA-SC

8. Secondary Outcome: Percentage of Participants With a Response in the Dysmenorrhea Component of the CPSSS Over Time
Description: The CPSSS consists of 5 components that address dysmenorrhea, dyspareunia, non-menstrual pelvic pain, pelvic tenderness, and pelvic induration. Each component was scored on a scale of 0 to 3 (0 = absent, 1 = mild, 2 = moderate, and 3 = severe). The dysmenorrhea score was based on the participant's response to the question "Have you had painful menstruation during the last 28 days?".
  Participants were classified as responders for dysmenorrhea if they reported a 1 point or greater reduction (improvement) from baseline.
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, 24, 28, 36, and 48
Population: All randomized participants who received at least one oral dose of study drug, an initial subcutaneous injection, and either reported at least 7 e-diary VAS values or provided an assessment of either dysmenorrhea or non-menstrual pelvic pain at week 4 or later during the treatment phase (intent-to-treat) with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 83
percentage of participants
  Week 4: number analyzed (Participants) | 81 | 83 | 83
  Week 4 | 75.3 | 80.7 | 74.7
  Week 8: number analyzed (Participants) | 75 | 75 | 73
  Week 8 | 84.0 | 84.0 | 79.5
  Week 12: number analyzed (Participants) | 71 | 73 | 67
  Week 12 | 73.2 | 82.2 | 82.1
  Week 16: number analyzed (Participants) | 64 | 69 | 57
  Week 16 | 87.5 | 82.6 | 91.2
  Week 20: number analyzed (Participants) | 60 | 68 | 54
  Week 20 | 81.7 | 76.5 | 83.3
  Week 24: number analyzed (Participants) | 57 | 65 | 51
  Week 24 | 86.0 | 73.8 | 86.3
  Week 28: number analyzed (Participants) | 48 | 61 | 45
  Week 28 | 70.8 | 57.4 | 93.3
  Week 36: number analyzed (Participants) | 40 | 56 | 41
  Week 36 | 52.5 | 44.6 | 80.5
  Week 48: number analyzed (Participants) | 33 | 55 | 39
  Week 48 | 63.6 | 58.2 | 66.7

9. Secondary Outcome: Percentage of Participants With a Response in the Non-menstrual Pelvic Pain Component of the CPSSS Over Time
Description: as for outcome 7
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, 24, 28, 36, and 48
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 83
percentage of participants
  Week 4: number analyzed (Participants) | 81 | 83 | 83
  Week 4 | 74.1 | 56.6 | 68.7
  Week 8: number analyzed (Participants) | 75 | 75 | 73
  Week 8 | 82.7 | 76.0 | 82.2
  Week 12: number analyzed (Participants) | 71 | 73 | 67
  Week 12 | 74.6 | 82.2 | 71.6
  Week 16: number analyzed (Participants) | 64 | 69 | 57
  Week 16 | 82.8 | 78.3 | 70.2
  Week 20: number analyzed (Participants) | 60 | 68 | 54
  Week 20 | 81.7 | 80.9 | 75.9
  Week 24: number analyzed (Participants) | 57 | 65 | 51
  Week 24 | 86.0 | 76.9 | 76.5
  Week 28: number analyzed (Participants) | 48 | 61 | 45
  Week 28 | 66.7 | 60.7 | 73.3
  Week 36: number analyzed (Participants) | 40 | 56 | 41
  Week 36 | 67.5 | 60.7 | 68.3
  Week 48: number analyzed (Participants) | 33 | 55 | 39
  Week 48 | 66.7 | 56.4 | 71.8

10. Secondary Outcome: Change From Baseline in Total CPSSS During the Treatment Period
Description: The CPSSS consists of 5 components that address dysmenorrhea, dyspareunia, non-menstrual pelvic pain, pelvic tenderness, and pelvic induration. Each component was scored on a scale of 0 to 3 (0 = absent, 1 = mild, 2 = moderate, and 3 = severe).
  Dysmenorrhea, dyspareunia, and nonmenstrual pelvic pain scores are based on the participant's assessment, pelvic tenderness and induration were assessed by the investigator based on findings associated with a pelvic examination.
  The total CPSSS has a maximum possible value of 15 (total score range: 0 to 15, where a lower score indicates less signs and symptoms of endometriosis or better functioning).
  Change from baseline was analyzed using a mixed-effects repeated measures (MERM) analysis of covariance model which included fixed effects for treatment, time, treatment-by-time interaction, a random effect for patient, and terms for baseline value and the baseline-by-time interaction.
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 83
units on a scale
  Week 4: number analyzed (Participants) | 81 | 83 | 81
  Week 4 | -3.9 (0.29) | -3.7 (0.29) | -3.8 (0.29)
  Week 8: number analyzed (Participants) | 74 | 75 | 73
  Week 8 | -4.9 (0.30) | -4.8 (0.30) | -4.5 (0.30)
  Week 12: number analyzed (Participants) | 70 | 72 | 67
  Week 12 | -4.6 (0.31) | -5.1 (0.30) | -4.2 (0.31)
  Week 16: number analyzed (Participants) | 64 | 69 | 56
  Week 16 | -5.5 (0.32) | -5.4 (0.31) | -4.6 (0.33)
  Week 20: number analyzed (Participants) | 60 | 68 | 54
  Week 20 | -5.1 (0.33) | -5.3 (0.31) | -4.8 (0.34)
  Week 24: number analyzed (Participants) | 57 | 64 | 50
  Week 24 | -5.5 (0.34) | -5.2 (0.32) | -5.3 (0.36)
Statistical Analysis 1: Comparison: Elagolix 150 mg QD; Within-group analysis of change from baseline in total CPSSS at week 24. Change from baseline was analyzed using a mixed-effects repeated measures (MERM) analysis of covariance model which included fixed effects for treatment, time, treatment-by-time interaction, a random effect for patient, and terms for baseline value and the baseline-by-time interaction; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -5.5, 95% CI 2-sided [-6.2 to -4.8]
Statistical Analysis 2: Comparison: Elagolix 75 mg BID; [analysis description as in outcome 10, analysis 1]; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -5.2, 95% CI 2-sided [-5.8 to -4.5]
Statistical Analysis 3: Comparison: DMPA-SC; [analysis description as in outcome 10, analysis 1]; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -5.3, 95% CI 2-sided [-6.0 to -4.6]

11. Secondary Outcome: Change From Baseline in Total CPSSS Excluding Dyspareunia During the Treatment Period
Description: The CPSSS consists of 5 components that address dysmenorrhea, dyspareunia, non-menstrual pelvic pain, pelvic tenderness, and pelvic induration. Each component was scored on a scale of 0 to 3 (0 = absent, 1 = mild, 2 = moderate, and 3 = severe).
  Dysmenorrhea, dyspareunia, and nonmenstrual pelvic pain scores are based on the participant's assessment, pelvic tenderness and induration were assessed by the investigator based on findings associated with a pelvic examination.
  The total CPSSS excluding dyspareunia has a maximum possible value of 12 (total score range: 0 to 12, where a lower score indicates less signs and symptoms of endometriosis or better functioning).
  Change from baseline was analyzed using a mixed-effects repeated measures (MERM) analysis of covariance model which included fixed effects for treatment, time, treatment-by-time interaction, a random effect for patient, and terms for baseline value and the baseline-by-time interaction.
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 83
units on a scale
  Week 4: number analyzed (Participants) | 81 | 83 | 81
  Week 4 | -3.4 (0.25) | -3.4 (0.25) | -3.3 (0.25)
  Week 8: number analyzed (Participants) | 74 | 75 | 73
  Week 8 | -4.1 (0.26) | -4.2 (0.26) | -3.8 (0.26)
  Week 12: number analyzed (Participants) | 70 | 72 | 67
  Week 12 | -3.8 (0.26) | -4.4 (0.26) | -3.7 (0.27)
  Week 16: number analyzed (Participants) | 64 | 69 | 56
  Week 16 | -4.6 (0.27) | -4.6 (0.27) | -3.9 (0.29)
  Week 20: number analyzed (Participants) | 60 | 68 | 54
  Week 20 | -4.4 (0.28) | -4.4 (0.27) | -4.1 (0.30)
  Week 24: number analyzed (Participants) | 57 | 64 | 50
  Week 24 | -4.6 (0.29) | -4.4 (0.28) | -4.5 (0.31)
Statistical Analysis 1: Comparison: Elagolix 150 mg QD; Within-group analysis of change from baseline in total CPSSS excluding dyspareunia at week 24. Change from baseline was analyzed using a mixed-effects repeated measures (MERM) analysis of covariance model which included fixed effects for treatment, time, treatment-by-time interaction, a random effect for patient, and terms for baseline value and the baseline-by-time interaction; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -4.6, 95% CI 2-sided [-5.1 to -4.0]
Statistical Analysis 2: Comparison: Elagolix 75 mg BID; [analysis description as in outcome 11, analysis 1]; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -4.4, 95% CI 2-sided [-5.0 to -3.9]
Statistical Analysis 3: Comparison: DMPA-SC; [analysis description as in outcome 11, analysis 1]; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -4.5, 95% CI 2-sided [-5.1 to -3.9]

12. Secondary Outcome: Change From Baseline in Dysmenorrhea Component of the CPSSS During the Treatment Period
Description: The CPSSS consists of 5 components that address dysmenorrhea, dyspareunia, non-menstrual pelvic pain, pelvic tenderness, and pelvic induration. Each component was scored on a scale of 0 to 3 (0 = absent, 1 = mild, 2 = moderate, and 3 = severe).
  The dysmenorrhea score was based on the participant's response to the question "Have you had painful menstruation during the last 28 days?".
  Change from baseline was analyzed using a mixed-effects repeated measures (MERM) analysis of covariance model which included fixed effects for treatment, time, treatment-by-time interaction, a random effect for patient, and terms for baseline value and the baseline-by-time interaction.
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 83
units on a scale
  Week 4: number analyzed (Participants) | 81 | 83 | 83
  Week 4 | -1.4 (0.11) | -1.5 (0.11) | -1.3 (0.11)
  Week 8: number analyzed (Participants) | 75 | 75 | 73
  Week 8 | -1.6 (0.11) | -1.7 (0.11) | -1.5 (0.12)
  Week 12: number analyzed (Participants) | 71 | 73 | 67
  Week 12 | -1.3 (0.12) | -1.7 (0.12) | -1.5 (0.12)
  Week 16: number analyzed (Participants) | 64 | 69 | 57
  Week 16 | -1.6 (0.12) | -1.8 (0.12) | -1.8 (0.13)
  Week 20: number analyzed (Participants) | 60 | 68 | 54
  Week 20 | -1.4 (0.13) | -1.5 (0.12) | -1.4 (0.13)
  Week 24: number analyzed (Participants) | 57 | 65 | 51
  Week 24 | -1.5 (0.13) | -1.4 (0.12) | -1.7 (0.14)
Statistical Analysis 1: Comparison: Elagolix 150 mg QD; Within-group analysis of change from baseline in dysmenorrhea at week 24. Change from baseline was analyzed using a mixed-effects repeated measures (MERM) analysis of covariance model which included fixed effects for treatment, time, treatment-by-time interaction, a random effect for patient, and terms for baseline value and the baseline-by-time interaction; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -1.5, 95% CI 2-sided [-1.7 to -1.2]
Statistical Analysis 2: Comparison: Elagolix 75 mg BID; [analysis description as in outcome 12, analysis 1]; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -1.4, 95% CI 2-sided [-1.6 to -1.2]
Statistical Analysis 3: Comparison: DMPA-SC; [analysis description as in outcome 12, analysis 1]; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -1.7, 95% CI 2-sided [-1.9 to -1.4]

13. Secondary Outcome: Change From Baseline in Dyspareunia Component of the CPSSS During the Treatment Period
Description: The CPSSS consists of 5 components that address dysmenorrhea, dyspareunia, non-menstrual pelvic pain, pelvic tenderness, and pelvic induration. Each component was scored on a scale of 0 to 3 (0 = absent, 1 = mild, 2 = moderate, and 3 = severe).
  The dyspareunia score was based on the participant's response to the question "Have you had painful intercourse during the last 28 days?" Change from baseline was analyzed using a mixed-effects repeated measures (MERM) analysis of covariance model which included fixed effects for treatment, time, treatment-by-time interaction, a random effect for patient, and terms for baseline value and the baseline-by-time interaction.
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 83
units on a scale
  Week 4: number analyzed (Participants) | 62 | 48 | 59
  Week 4 | -0.6 (0.11) | -0.4 (0.13) | -0.5 (0.11)
  Week 8: number analyzed (Participants) | 53 | 47 | 51
  Week 8 | -0.9 (0.12) | -0.7 (0.13) | -0.8 (0.12)
  Week 12: number analyzed (Participants) | 51 | 46 | 49
  Week 12 | -1.0 (0.12) | -0.8 (0.13) | -0.6 (0.12)
  Week 16: number analyzed (Participants) | 45 | 42 | 35
  Week 16 | -1.2 (0.13) | -1.0 (0.13) | -0.8 (0.14)
  Week 20: number analyzed (Participants) | 41 | 38 | 33
  Week 20 | -0.9 (0.13) | -1.0 (0.14) | -0.8 (0.14)
  Week 24: number analyzed (Participants) | 39 | 38 | 30
  Week 24 | -1.2 (0.13) | -1.0 (0.14) | -0.8 (0.15)
Statistical Analysis 1: Comparison: Elagolix 150 mg QD; Within-group analysis of change from baseline in dyspareunia at week 24. Change from baseline was analyzed using a mixed-effects repeated measures (MERM) analysis of covariance model which included fixed effects for treatment, time, treatment-by-time interaction, a random effect for patient, and terms for baseline value and the baseline-by-time interaction; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -1.2, 95% CI 2-sided [-1.4 to -0.9]
Statistical Analysis 2: Comparison: Elagolix 75 mg BID; [analysis description as in outcome 13, analysis 1]; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -1.0, 2% CI 2-sided [-1.2 to -0.7]
Statistical Analysis 3: Comparison: DMPA-SC; [analysis description as in outcome 13, analysis 1]; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -0.8, 95% CI 2-sided [-1.1 to -0.5]

14. Secondary Outcome: Change From Baseline in Non-menstrual Pelvic Pain Component of the CPSSS During the Treatment Period
Description: The CPSSS consists of 5 components that address dysmenorrhea, dyspareunia, non-menstrual pelvic pain, pelvic tenderness, and pelvic induration. Each component was scored on a scale of 0 to 3 (0 = absent, 1 = mild, 2 = moderate, and 3 = severe).
  The non-menstrual pelvic pain score was based on participant's response to the question "Have you had pelvic pain during the last 28 days?".
  Change from baseline was analyzed using a mixed-effects repeated measures (MERM) analysis of covariance model which included fixed effects for treatment, time, treatment-by-time interaction, a random effect for patient, and terms for baseline value and the baseline-by-time interaction.
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 83
units on a scale
  Week 4: number analyzed (Participants) | 81 | 83 | 83
  Week 4 | -0.9 (0.09) | -0.8 (0.09) | -0.8 (0.09)
  Week 8: number analyzed (Participants) | 75 | 75 | 73
  Week 8 | -1.1 (0.09) | -1.1 (0.09) | -1.1 (0.09)
  Week 12: number analyzed (Participants) | 71 | 73 | 67
  Week 12 | -1.0 (0.09) | -1.1 (0.09) | -0.9 (0.10)
  Week 16: number analyzed (Participants) | 64 | 69 | 57
  Week 16 | -1.2 (0.10) | -1.2 (0.09) | -0.9 (0.10)
  Week 20: number analyzed (Participants) | 60 | 68 | 54
  Week 20 | -1.1 (0.10) | -1.3 (0.10) | -1.0 (0.11)
  Week 24: number analyzed (Participants) | 57 | 65 | 51
  Week 24 | -1.2 (0.10) | -1.2 (0.10) | -1.1 (0.11)
Statistical Analysis 1: Comparison: Elagolix 150 mg QD; Within-group analysis of change from baseline in non-menstrual pelvic pain at week 24. Change from baseline was analyzed using a mixed-effects repeated measures (MERM) analysis of covariance model which included fixed effects for treatment, time, treatment-by-time interaction, a random effect for patient, and terms for baseline value and the baseline-by-time interaction; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -1.2, 95% CI 2-sided [-1.4 to -1.0]
Statistical Analysis 2: Comparison: Elagolix 75 mg BID; [analysis description as in outcome 14, analysis 1]; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -1.2, 95% CI 2-sided [-1.4 to -1.0]
Statistical Analysis 3: Comparison: DMPA-SC; [analysis description as in outcome 14, analysis 1]; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -1.1, 95% CI 2-sided [-1.3 to -0.8]

15. Secondary Outcome: Change From Baseline in Pelvic Tenderness Component of the CPSSS During the Treatment Period
Description: The CPSSS consists of 5 components that address dysmenorrhea, dyspareunia, non-menstrual pelvic pain, pelvic tenderness, and pelvic induration. Each component was scored on a scale of 0 to 3 (0 = absent, 1 = mild, 2 = moderate, and 3 = severe).
  Pelvic tenderness was assessed by the investigator based on findings associated with a pelvic examination.
  Change from baseline was analyzed using a mixed-effects repeated measures (MERM) analysis of covariance model which included fixed effects for treatment, time, treatment-by-time interaction, a random effect for patient, and terms for baseline value and the baseline-by-time interaction.
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 83
units on a scale
  Week 4: number analyzed (Participants) | 81 | 83 | 81
  Week 4 | -0.6 (0.08) | -0.7 (0.08) | -0.7 (0.08)
  Week 8: number analyzed (Participants) | 74 | 75 | 73
  Week 8 | -0.8 (0.09) | -0.8 (0.08) | -0.7 (0.09)
  Week 12: number analyzed (Participants) | 70 | 72 | 67
  Week 12 | -0.8 (0.09) | -0.9 (0.09) | -0.7 (0.09)
  Week 16: number analyzed (Participants) | 64 | 69 | 56
  Week 16 | -1.0 (0.09) | -0.9 (0.09) | -0.6 (0.09)
  Week 20: number analyzed (Participants) | 60 | 68 | 54
  Week 20 | -1.0 (0.09) | -0.8 (0.09) | -0.9 (0.10)
  Week 24: number analyzed (Participants) | 57 | 64 | 50
  Week 24 | -1.0 (0.09) | -1.0 (0.09) | -0.9 (0.10)
Statistical Analysis 1: Comparison: Elagolix 150 mg QD; Within-group analysis of change from baseline in pelvic tenderness at week 24. Change from baseline was analyzed using a mixed-effects repeated measures (MERM) analysis of covariance model which included fixed effects for treatment, time, treatment-by-time interaction, a random effect for patient, and terms for baseline value and the baseline-by-time interaction; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -1.0, 95% CI 2-sided [-1.2 to -0.8]
Statistical Analysis 2: Comparison: Elagolix 75 mg BID; [analysis description as in outcome 15, analysis 1]; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -1.0, 95% CI 2-sided [-1.1 to -0.8]
Statistical Analysis 3: Comparison: DMPA-SC; [analysis description as in outcome 15, analysis 1]; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -0.9, 95% CI 2-sided [-1.1 to -0.7]

16. Secondary Outcome: Change From Baseline in Pelvic Induration Component of the CPSSS During the Treatment Period
Description: The CPSSS consists of 5 components that address dysmenorrhea, dyspareunia, non-menstrual pelvic pain, pelvic tenderness, and pelvic induration. Each component was scored on a scale of 0 to 3 (0 = absent, 1 = mild, 2 = moderate, and 3 = severe).
  Pelvic induration was assessed by the investigator based on findings associated with a pelvic examination.
  Change from baseline was analyzed using a mixed-effects repeated measures (MERM) analysis of covariance model which included fixed effects for treatment, time, treatment-by-time interaction, a random effect for patient, and terms for baseline value and the baseline-by-time interaction.
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 83
units on a scale
  Week 4: number analyzed (Participants) | 81 | 83 | 81
  Week 4 | -0.4 (0.08) | -0.5 (0.08) | -0.5 (0.08)
  Week 8: number analyzed (Participants) | 74 | 75 | 73
  Week 8 | -0.7 (0.08) | -0.6 (0.08) | -0.6 (0.08)
  Week 12: number analyzed (Participants) | 70 | 72 | 67
  Week 12 | -0.7 (0.08) | -0.8 (0.08) | -0.6 (0.08)
  Week 16: number analyzed (Participants) | 64 | 69 | 56
  Week 16 | -0.9 (0.09) | -0.8 (0.08) | -0.7 (0.09)
  Week 20: number analyzed (Participants) | 60 | 68 | 54
  Week 20 | -0.9 (0.09) | -0.8 (0.08) | -0.8 (0.09)
  Week 24: number analyzed (Participants) | 57 | 64 | 50
  Week 24 | -0.9 (0.09) | -0.9 (0.09) | -0.8 (0.10)
Statistical Analysis 1: Comparison: Elagolix 150 mg QD; Within-group analysis of change from baseline in pelvic induration at week 24. Change from baseline was analyzed using a mixed-effects repeated measures (MERM) analysis of covariance model which included fixed effects for treatment, time, treatment-by-time interaction, a random effect for patient, and terms for baseline value and the baseline-by-time interaction; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -0.9, 95% CI 2-sided [-1.0 to -0.7]
Statistical Analysis 2: Comparison: Elagolix 75 mg BID; [analysis description as in outcome 16, analysis 1]; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -0.9, 95% CI 2-sided [-1.1 to -0.7]
Statistical Analysis 3: Comparison: DMPA-SC; [analysis description as in outcome 16, analysis 1]; Test type: Other; p < 0.0001, t-test, 2 sided; Least squares mean = -0.8, 95% CI 2-sided [-0.9 to -0.6]

17. Secondary Outcome: Change From Baseline in in Monthly Peak Visual Analog Scale (VAS) for Pelvic Pain
Description: The VAS for pelvic pain was used as an assessment of pain intensity. The VAS was a horizontal line on which the left extreme was labeled "no pain" and the right extreme was labeled "worst pain ever felt" scored on a scale from of 0 (no pain) to 100 (worst pain ever felt). Participants indicated the worst level of pain felt over a 24-hour period by ''ticking'' the horizontal line on their e-Diary at approximately the same time each day. Monthly peak VAS for pelvic pain was defined as the maximum VAS pain score reported for an individual participant from the previous visit to the day of the current scheduled visit.
  Change from baseline was analyzed using a mixed-effects repeated measures (MERM) analysis of covariance model which included fixed effects for treatment, time, treatment-by-time interaction, a random effect for patient, and terms for baseline value and the baseline-by-time interaction.
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 83
units on a scale
  Week 4: number analyzed (Participants) | 83 | 84 | 82
  Week 4 | -18.2 (2.97) | -14.4 (2.96) | -15.4 (2.98)
  Week 8: number analyzed (Participants) | 76 | 78 | 74
  Week 8 | -26.3 (3.06) | -28.1 (3.02) | -27.1 (3.08)
  Week 12: number analyzed (Participants) | 70 | 73 | 66
  Week 12 | -31.3 (3.14) | -32.7 (3.09) | -24.9 (3.20)
  Week 16: number analyzed (Participants) | 65 | 67 | 58
  Week 16 | -32.1 (3.24) | -37.8 (3.19) | -30.8 (3.38)
  Week 20: number analyzed (Participants) | 58 | 66 | 54
  Week 20 | -29.0 (3.40) | -37.9 (3.23) | -31.0 (3.51)
  Week 24: number analyzed (Participants) | 55 | 63 | 50
  Week 24 | -32.3 (3.51) | -32.9 (3.31) | -35.8 (3.65)
Statistical Analysis 1: Comparison: Elagolix 150 mg QD; Within-group analysis of change from baseline in peak VAS for pelvic pain at week 24. Change from baseline was analyzed using a mixed-effects repeated measures (MERM) analysis of covariance model which included fixed effects for treatment, time, treatment-by-time interaction, a random effect for patient, and terms for baseline value and the baseline-by-time interaction; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -32.3, 95% CI 2-sided [-39.2 to -25.4]
Statistical Analysis 2: Comparison: Elagolix 75 mg BID; [analysis description as in outcome 17, analysis 1]; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -32.9, 95% CI 2-sided [-39.4 to -26.4]
Statistical Analysis 3: Comparison: DMPA-SC; [analysis description as in outcome 17, analysis 1]; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -35.8, 95% CI 2-sided [-43.0 to -28.6]

18. Secondary Outcome: Change From Baseline in in Monthly Mean Visual Analog Scale (VAS) for Pelvic Pain
Description: The VAS for pelvic pain was used as an assessment of pain intensity. The VAS was a horizontal line on which the left extreme was labeled "no pain" and the right extreme was labeled "worst pain ever felt" scored on a scale from of 0 (no pain) to 100 (worst pain ever felt). Participants indicated the worst level of pain felt over a 24-hour period by ''ticking'' the horizontal line on their e-Diary at approximately the same time each day. Monthly mean VAS for pelvic pain defined as the average of all VAS pain scores reported for an individual participant from the previous visit to the day of the current scheduled visit.
  Change from baseline was analyzed using a mixed-effects repeated measures (MERM) analysis of covariance model which included fixed effects for treatment, time, treatment-by-time interaction, a random effect for patient, and terms for baseline value and the baseline-by-time interaction.
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 83
units on a scale
  Week 4: number analyzed (Participants) | 83 | 84 | 82
  Week 4 | -10.2 (1.59) | -11.7 (1.58) | -10.2 (1.59)
  Week 8: number analyzed (Participants) | 76 | 78 | 74
  Week 8 | -14.0 (2.09) | -17.8 (2.06) | -15.9 (2.10)
  Week 12: number analyzed (Participants) | 70 | 73 | 66
  Week 12 | -17.7 (2.24) | -23.4 (2.19) | -15.5 (2.27)
  Week 16: number analyzed (Participants) | 65 | 67 | 58
  Week 16 | -17.8 (2.51) | -23.6 (2.45) | -17.3 (2.57)
  Week 20: number analyzed (Participants) | 58 | 66 | 54
  Week 20 | -16.6 (2.53) | -24.1 (2.43) | -17.1 (2.59)
  Week 24: number analyzed (Participants) | 55 | 63 | 50
  Week 24 | -18.2 (2.57) | -23.4 (2.47) | -17.9 (2.64)
Statistical Analysis 1: Comparison: Elagolix 150 mg QD; Within-group analysis of change from baseline in monthly mean VAS for pelvic pain at week 24. Change from baseline was analyzed using a mixed-effects repeated measures (MERM) analysis of covariance model which included fixed effects for treatment, time, treatment-by-time interaction, a random effect for patient, and terms for baseline value and the baseline-by-time interaction; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -18.2, 95% CI 2-sided [-23.3 to -13.1]
Statistical Analysis 2: Comparison: Elagolix 75 mg BID; [analysis description as in outcome 18, analysis 1]; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -23.4, 95% CI 2-sided [-28.3 to -18.5]
Statistical Analysis 3: Comparison: DMPA-SC; [analysis description as in outcome 17, analysis 1]; Test type: Other; p < 0.0001, t-test, 2 sided — P-value for test of null hypothesis that the treatment group least squares mean is equal to zero; Least squares mean = -17.9, 95% CI 2-sided [-23.1 to -12.7]

19. Secondary Outcome: Change From Baseline in Endometriosis Health Profile-5 (EHP-5) Pain Dimension
Description: The EHP-5 is an instrument to measure health-related quality of life in women with endometriosis. The EHP-5 consists of two parts:
  * A core questionnaire consisting of five questions that measure the areas of pain, control and powerlessness, emotional well-being, social support, and self-image
  * A supplemental questionnaire consisting of six additional questions, five of which were recorded in this study: work, relationship with children, sexual intercourse, feelings about the medical profession and treatment.
  Each question was scored on a five point scale (Never = 0, Rarely = 25, Sometimes = 50, Often = 75, Always = 100), where 0 indicates the best health status and 100 worst health status. A negative change from baseline score indicates improvement in quality of life.
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 83
units on a scale
  Week 4: number analyzed (Participants) | 81 | 82 | 83
  Week 4 | -20.7 (2.4) | -22.9 (2.6) | -18.7 (2.5)
  Week 8: number analyzed (Participants) | 74 | 75 | 73
  Week 8 | -22.0 (3.1) | -30.0 (2.5) | -24.3 (2.6)
  Week 12: number analyzed (Participants) | 71 | 73 | 67
  Week 12 | -23.2 (3.1) | -28.4 (3.2) | -25.4 (3.4)
  Week 16: number analyzed (Participants) | 64 | 69 | 57
  Week 16 | -30.9 (3.1) | -31.9 (2.8) | -29.8 (3.7)
  Week 20: number analyzed (Participants) | 60 | 68 | 53
  Week 20 | -26.3 (3.8) | -29.8 (2.8) | -28.3 (3.6)
  Week 24: number analyzed (Participants) | 57 | 65 | 51
  Week 24 | -28.9 (3.2) | -28.5 (3.2) | -30.9 (4.1)

20. Secondary Outcome: Change From Baseline in EHP-5 Control and Powerlessness Dimension
Description: as for outcome 19
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 83
units on a scale
  Week 4: number analyzed (Participants) | 81 | 82 | 83
  Week 4 | -19.8 (2.9) | -24.7 (3.0) | -22.9 (2.6)
  Week 8: number analyzed (Participants) | 74 | 75 | 73
  Week 8 | -27.7 (3.1) | -33.0 (3.5) | -31.2 (3.5)
  Week 12: number analyzed (Participants) | 71 | 73 | 67
  Week 12 | -30.6 (3.3) | -31.2 (3.8) | -26.1 (4.0)
  Week 16: number analyzed (Participants) | 64 | 69 | 57
  Week 16 | -34.4 (3.7) | -33.3 (3.8) | -31.1 (4.3)
  Week 20: number analyzed (Participants) | 60 | 68 | 53
  Week 20 | -32.9 (3.8) | -33.1 (4.2) | -34.9 (4.4)
  Week 24: number analyzed (Participants) | 57 | 65 | 51
  Week 24 | -37.3 (3.8) | -33.1 (3.8) | -35.8 (5.0)

21. Secondary Outcome: Change From Baseline in EHP-5 Emotional Well-being Dimension
Description: as for outcome 19
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 83
units on a scale
  Week 4: number analyzed (Participants) | 81 | 82 | 83
  Week 4 | -12.7 (2.5) | -10.4 (2.7) | -5.1 (2.8)
  Week 8: number analyzed (Participants) | 74 | 75 | 73
  Week 8 | -20.6 (2.7) | -16.0 (3.1) | -13.4 (2.9)
  Week 12: number analyzed (Participants) | 71 | 73 | 67
  Week 12 | -18.0 (3.0) | -21.9 (3.2) | -14.6 (2.6)
  Week 16: number analyzed (Participants) | 64 | 69 | 57
  Week 16 | -21.1 (3.3) | -20.7 (3.6) | -14.9 (3.7)
  Week 20: number analyzed (Participants) | 60 | 68 | 53
  Week 20 | -20.8 (3.7) | -22.8 (3.1) | -18.4 (3.8)
  Week 24: number analyzed (Participants) | 57 | 65 | 51
  Week 24 | -24.1 (3.6) | -23.8 (3.4) | -25.5 (4.2)

22. Secondary Outcome: Change From Baseline in EHP-5 Social Support Dimension
Description: as for outcome 19
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 83
units on a scale
  Week 4: number analyzed (Participants) | 81 | 82 | 83
  Week 4 | -25.3 (3.0) | -26.5 (3.4) | -19.6 (2.9)
  Week 8: number analyzed (Participants) | 74 | 75 | 73
  Week 8 | -31.4 (3.5) | -33.7 (3.9) | -29.8 (3.4)
  Week 12: number analyzed (Participants) | 70 | 73 | 67
  Week 12 | -36.8 (3.7) | -34.6 (4.4) | -28.4 (3.6)
  Week 16: number analyzed (Participants) | 64 | 69 | 57
  Week 16 | -42.2 (4.0) | -37.0 (4.3) | -32.0 (3.7)
  Week 20: number analyzed (Participants) | 60 | 68 | 53
  Week 20 | -42.1 (4.2) | -39.0 (4.4) | -34.9 (3.9)
  Week 24: number analyzed (Participants) | 57 | 65 | 51
  Week 24 | -43.4 (4.1) | -40.0 (4.4) | -32.8 (5.1)

23. Secondary Outcome: Change From Baseline in EHP-5 Self Image Dimension
Description: as for outcome 19
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 83
units on a scale
  Week 4: number analyzed (Participants) | 81 | 82 | 83
  Week 4 | -11.1 (3.3) | -20.1 (2.9) | -11.1 (3.5)
  Week 8: number analyzed (Participants) | 74 | 75 | 73
  Week 8 | -19.6 (3.3) | -22.7 (3.3) | -17.5 (3.8)
  Week 12: number analyzed (Participants) | 71 | 73 | 67
  Week 12 | -21.1 (4.0) | -22.6 (3.2) | -18.3 (4.1)
  Week 16: number analyzed (Participants) | 64 | 69 | 57
  Week 16 | -20.3 (3.6) | -25.7 (3.1) | -18.9 (3.9)
  Week 20: number analyzed (Participants) | 60 | 68 | 53
  Week 20 | -20.8 (4.3) | -26.1 (3.4) | -19.3 (4.4)
  Week 24: number analyzed (Participants) | 57 | 65 | 51
  Week 24 | -23.7 (4.1) | -26.9 (3.8) | -24.5 (4.9)

24. Secondary Outcome: Change From Baseline in EHP-5 Work Dimension
Description: The EHP-5 is an instrument to measure health-related quality of life in women with endometriosis. The EHP-5 consists of two parts:
  * A core questionnaire consisting of five questions that measure the areas of pain, control and powerlessness, emotional well-being, social support, and self-image
  * A supplemental questionnaire consisting of six additional questions, five of which were recorded in this study: work, relationship with children, sexual intercourse, feelings about the medical profession and treatment.
  Each question was scored on a five point scale (Never = 0, Rarely = 25, Sometimes = 50, Often = 75, Always = 100), or Not Relevant (no score), where 0 indicates the best health status and 100 worst health status. A negative change from baseline score indicates improvement in quality of life.
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 83
units on a scale
  Week 4: number analyzed (Participants) | 73 | 73 | 75
  Week 4 | -20.5 (3.2) | -20.9 (2.8) | -21.0 (2.6)
  Week 8: number analyzed (Participants) | 66 | 66 | 64
  Week 8 | -21.2 (3.5) | -25.8 (3.1) | -25.8 (3.3)
  Week 12: number analyzed (Participants) | 62 | 66 | 58
  Week 12 | -21.8 (3.8) | -24.2 (3.3) | -25.4 (3.7)
  Week 16: number analyzed (Participants) | 58 | 63 | 47
  Week 16 | -24.6 (3.9) | -26.6 (3.2) | -26.6 (4.0)
  Week 20: number analyzed (Participants) | 54 | 61 | 45
  Week 20 | -24.1 (4.2) | -27.5 (3.1) | -29.4 (4.1)
  Week 24: number analyzed (Participants) | 51 | 58 | 44
  Week 24 | -24.0 (4.0) | -26.7 (3.1) | -27.8 (4.2)

25. Secondary Outcome: Change From Baseline in EHP-5 Relationship With Children Dimension
Description: as for outcome 24
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 83
units on a scale
  Week 4: number analyzed (Participants) | 42 | 37 | 45
  Week 4 | -16.1 (4.4) | -18.9 (3.8) | -16.1 (3.9)
  Week 8: number analyzed (Participants) | 39 | 36 | 39
  Week 8 | -19.9 (4.5) | -20.8 (3.8) | -24.4 (3.9)
  Week 12: number analyzed (Participants) | 37 | 35 | 35
  Week 12 | -23.0 (4.8) | -20.7 (4.2) | -28.6 (4.8)
  Week 16: number analyzed (Participants) | 31 | 32 | 30
  Week 16 | -24.2 (4.7) | -26.6 (4.2) | -25.8 (5.0)
  Week 20: number analyzed (Participants) | 27 | 28 | 28
  Week 20 | -27.8 (4.3) | -25.0 (4.1) | -28.6 (5.7)
  Week 24: number analyzed (Participants) | 26 | 29 | 26
  Week 24 | -29.8 (4.6) | -23.3 (4.3) | -31.7 (6.0)

26. Secondary Outcome: Change From Baseline in EHP-5 Intercourse Dimension
Description: as for outcome 24
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 83
units on a scale
  Week 4: number analyzed (Participants) | 71 | 65 | 69
  Week 4 | -17.3 (3.3) | -18.5 (3.6) | -17.4 (3.3)
  Week 8: number analyzed (Participants) | 62 | 57 | 61
  Week 8 | -25.8 (3.5) | -27.2 (3.8) | -20.5 (4.3)
  Week 12: number analyzed (Participants) | 61 | 56 | 55
  Week 12 | -29.1 (3.7) | -29.5 (4.0) | -20.5 (4.4)
  Week 16: number analyzed (Participants) | 52 | 54 | 43
  Week 16 | -31.7 (4.3) | -29.2 (3.8) | -23.3 (5.1)
  Week 20: number analyzed (Participants) | 48 | 52 | 41
  Week 20 | -30.7 (4.4) | -31.7 (4.2) | -25.0 (5.2)
  Week 24: number analyzed (Participants) | 46 | 45 | 39
  Week 24 | -35.3 (4.4) | -33.9 (4.4) | -29.5 (5.4)

27. Secondary Outcome: Change From Baseline in EHP-5 Medical Profession Dimension
Description: as for outcome 24
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 83
units on a scale
  Week 4: number analyzed (Participants) | 70 | 69 | 71
  Week 4 | -13.2 (3.4) | -9.1 (2.6) | -12.0 (2.6)
  Week 8: number analyzed (Participants) | 62 | 63 | 65
  Week 8 | -15.3 (3.0) | -14.7 (3.2) | -13.5 (3.2)
  Week 12: number analyzed (Participants) | 60 | 60 | 60
  Week 12 | -16.7 (3.4) | -14.2 (3.7) | -15.0 (3.2)
  Week 16: number analyzed (Participants) | 53 | 59 | 49
  Week 16 | -18.9 (3.6) | -14.4 (3.4) | -17.9 (3.5)
  Week 20: number analyzed (Participants) | 48 | 60 | 48
  Week 20 | -18.2 (3.8) | -14.6 (3.2) | -15.6 (3.8)
  Week 24: number analyzed (Participants) | 48 | 57 | 47
  Week 24 | -18.8 (3.5) | -14.0 (3.5) | -16.0 (4.1)

28. Secondary Outcome: Change From Baseline in EHP-5 Treatment Dimension
Description: as for outcome 24
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 83
units on a scale
  Week 4: number analyzed (Participants) | 52 | 53 | 55
  Week 4 | -27.4 (5.1) | -30.2 (4.5) | -26.8 (4.4)
  Week 8: number analyzed (Participants) | 48 | 50 | 47
  Week 8 | -32.8 (6.3) | -37.0 (4.8) | -29.8 (4.8)
  Week 12: number analyzed (Participants) | 45 | 45 | 42
  Week 12 | -35.0 (6.0) | -37.2 (5.5) | -28.0 (5.3)
  Week 16: number analyzed (Participants) | 38 | 47 | 35
  Week 16 | -36.8 (6.9) | -38.3 (4.6) | -28.6 (6.4)
  Week 20: number analyzed (Participants) | 35 | 46 | 33
  Week 20 | -35.7 (6.6) | -34.8 (5.2) | -35.6 (6.3)
  Week 24: number analyzed (Participants) | 33 | 42 | 32
  Week 24 | -35.6 (7.1) | -39.3 (5.0) | -28.9 (7.3)

29. Secondary Outcome: Percentage of Participants Using Analgesics During the Treatment Phase
Description: Analgesic use was collected as part of concomitant medications on a case report form that was administered at each scheduled visit.
Time Frame: 24 weeks
Population: All randomized participants who received at least one oral dose of study drug, an initial subcutaneous injection, and either reported at least 7 e-diary VAS values or provided an assessment of either dysmenorrhea or non-menstrual pelvic pain at week 4 or later during the treatment phase (intent-to-treat).
Measure: Number; unit: percentage of participants
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
Number analyzed (Participants) | 84 | 84 | 83
percentage of participants
  Antiinflammatory/Antirheumatics, Non-Steroids | 65.5 | 64.3 | 68.7
  Opioids | 23.8 | 25.0 | 33.7
  Other Analgesics and Antipyretics | 45.2 | 46.4 | 34.9

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 24 weeks after last dose (48 weeks)
Arm/Group | Elagolix 150 mg QD | Elagolix 75 mg BID | DMPA-SC
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/84 | 0/84
Serious Adverse Events (participants affected / at risk) | 3/84 | 3/84 | 6/84
Other Adverse Events (participants affected / at risk) | 63/84 | 59/84 | 63/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elagolix 150 mg QD (N=84) | Elagolix 75 mg BID (N=84) | DMPA-SC (N=84)
FOOD POISONING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
OVARIAN DYSGERMINOMA STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
DEPRESSION SUICIDAL (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
PELVIC CONGESTION (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
PELVIC PAIN (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elagolix 150 mg QD (N=84) | Elagolix 75 mg BID (N=84) | DMPA-SC (N=84)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 (2) | 0 (0) | 6 (7)
DIARRHOEA (Gastrointestinal disorders) | 4 (4) | 9 (10) | 8 (10)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 5 (7) | 3 (3)
NAUSEA (Gastrointestinal disorders) | 16 (21) | 13 (16) | 13 (20)
FATIGUE (General disorders) | 5 (5) | 3 (3) | 6 (6)
INFLUENZA (Infections and infestations) | 7 (7) | 5 (5) | 2 (2)
NASOPHARYNGITIS (Infections and infestations) | 9 (9) | 18 (22) | 9 (11)
SINUSITIS (Infections and infestations) | 7 (8) | 7 (12) | 6 (6)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 (10) | 10 (14) | 10 (10)
URINARY TRACT INFECTION (Infections and infestations) | 5 (6) | 8 (10) | 5 (5)
VAGINAL MYCOSIS (Infections and infestations) | 5 (6) | 4 (5) | 3 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (10) | 9 (13) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 (7) | 10 (11) | 4 (4)
DIZZINESS (Nervous system disorders) | 3 (4) | 6 (8) | 8 (9)
HEADACHE (Nervous system disorders) | 22 (48) | 23 (66) | 15 (64)
MIGRAINE (Nervous system disorders) | 4 (8) | 3 (3) | 5 (6)
ANXIETY (Psychiatric disorders) | 6 (6) | 4 (4) | 4 (4)
DEPRESSION (Psychiatric disorders) | 3 (3) | 6 (6) | 4 (4)
INSOMNIA (Psychiatric disorders) | 4 (4) | 7 (11) | 4 (4)
MOOD SWINGS (Psychiatric disorders) | 7 (8) | 6 (6) | 10 (10)
OVARIAN CYST (Reproductive system and breast disorders) | 5 (5) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7) | 3 (3)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 6 (6) | 3 (3)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 7 (8) | 3 (3)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (6) | 5 (5)
ACNE (Skin and subcutaneous tissue disorders) | 7 (7) | 2 (2) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.